CLINICAL TRIAL: NCT03581695
Title: Inflammatory Biomarkers of Pediatric Pulmonary Hypertension: a Prospective Cohort Study
Brief Title: Inflammatory Biomarkers of Pediatric Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Katherine Taylor, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000058900
Record Dates: First submitted 2018-06-20; First posted 2018-07-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary Hypertension and Congenital Heart Disease: Pulmonary Hypertension and Congenital Heart Disease
  Interventions: Other: Blood test
- Congenital Heart Disease: Congenital Heart Disease
  Interventions: Other: Blood test
- Healthy Controls: Healthy Controls
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood test

SUMMARY:
To investigate if the inflammatory protein, high mobility group box 1 (HMGB1), along with other inflammatory mediators, is elevated in pediatric patients with congenital heart disease (CHD) and pulmonary hypertension as compared to those with CHD alone, or with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

-patients of any age with congenital cardiac disease coming for catheterization of the right heart, or both the right and left heart.

Exclusion Criteria:

* active systemic infection
* current active cancer
* active cancer treatment
* prior bone marrow transplant
* prior solid organ transplant

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients of any age coming for cardiac catheterization and healthy controls coming for urology surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of HGMB1 | 1 day
  Measurement of HGMB1

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Taylor, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No